CLINICAL TRIAL: NCT00091156
Title: A Randomized Phase III Study of Follow Up With or Without Adjuvant Gefitinib (Iressa™) Following Chemotherapy in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Gefitinib After Chemotherapy in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: EORTC-08021; EORTC-08021; ILCP-01/03; 2004-001331-36 (EudraCT Number)
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: gefitinib
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. It is not yet known whether giving gefitinib after initial chemotherapy is effective in delaying the recurrence of non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying gefitinib to see how well it works compared to placebo in delaying tumor recurrence in patients who have undergone initial chemotherapy for stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall survival of patients with stage IIIB or IV non-small cell lung cancer that did not progress on prior first-line palliative induction chemotherapy when treated with adjuvant gefitinib vs placebo.

Secondary

* Compare progression-free survival of patients treated with these regimens.
* Determine the safety and toxicity of gefitinib in these patients.

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are stratified according to initial disease stage (IIIB vs IV), WHO performance status at the end of prior first-line palliative induction chemotherapy (0-1 vs 2), best patient response to prior first-line palliative induction chemotherapy (objective response vs stable disease), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral gefitinib once daily.
* Arm II: Patients receive oral placebo once daily. In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 598 patients (299 per treatment arm) will be accrued for this study within 8.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer meeting 1 of the following stage criteria:

  * Stage IIIB

    * Pleural fluid and/or supraclavicular nodes allowed provided patient is not eligible for consolidation radiotherapy
  * Stage IV disease
* No disease progression after 2-6 courses of prior platinum-containing first-line palliative induction chemotherapy
* Brain metastases allowed provided patients are asymptomatic after cranial irradiation completed at least 4 weeks ago

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Pulmonary

* No history, signs, or symptoms of clinically active interstitial lung disease

  * Patients with chronic, stable, asymptomatic radiographic changes are eligible

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up
* No other malignant disease within the past 5 years except basal cell skin cancer or adequately treated superficial carcinoma of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy (alopecia allowed)
* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Other

* No prior epidermal growth factor receptor inhibitors
* No concurrent administration of any of the following drugs:

  * Phenytoin
  * Carbamazepine
  * Rifampin
  * Phenobarbital
  * Hypericum perforatum (St. John's wort)
* No other concurrent anticancer therapy
* No other concurrent experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Estimated)
Dates: Start 2004-05; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Progression-free survival
Toxicity as assessed by CTC

CONTACTS AND LOCATIONS:
Overall Officials: Jan P. Van Meerbeeck, MD, PhD, Study Chair — University Ghent
Locations (28):
- Belgium (4):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Ghent University, Ghent
  - CHR - Clinique Saint Joseph - Hopital de Warqueguies, Mons
  - Clinique Sainte Elisabeth, Namur
- Bank Of Cyprus Oncology Centre, Nicosia, Cyprus
- National Cancer Institute of Egypt, Cairo, Egypt
- Italy (17):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale Santa Croce, Cuneo
  - Universita di Ferrara, Ferrara
  - Presidio Ospedaliero di Livorno, Livorno
  - Ospedale Luigi Sacco, Milan
  - Ospedale Niguarda Ca'Granda, Milan
  - Azienda Ospedaliera - Universitaria di Modena, Modena
  - Azienda Ospedaliera Maggiore Della Carita, Novara
  - Azienda Ospedale S. Luigi at University of Torino, Orbassano
  - Azienda Ospedaliera Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliera Di Parma, Parma
  - Azienda Ospedaliera "Santa Maria Degli Angeli", Pordenone
  - Ospedale Sta. Maria Delle Croci, Ravenna
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Azienda Ospedaliera S. Camillo-Forlanini, Rome
  - Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedale Civile Maggiore - Borgo Trento, Verona
- Netherlands (5):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Rijnstate Hospital, Arnhem
  - Kennemer Gasthuis - Locatie EG, Haarlem
  - Leiden University Medical Center, Leiden
  - St. Franciscus Gasthuis, Rotterdam

REFERENCES:
- [Result] Gaafar RM, Surmont VF, Scagliotti GV, Van Klaveren RJ, Papamichael D, Welch JJ, Hasan B, Torri V, van Meerbeeck JP; EORTC Lung Cancer Group and the Italian Lung Cancer Project. A double-blind, randomised, placebo-controlled phase III intergroup study of gefitinib in patients with advanced NSCLC, non-progressing after first line platinum-based chemotherapy (EORTC 08021/ILCP 01/03). Eur J Cancer. 2011 Oct;47(15):2331-40. doi: 10.1016/j.ejca.2011.06.045. Epub 2011 Jul 28. PMID 21802939